CLINICAL TRIAL: NCT04870645
Title: Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery
Brief Title: Advanced MRI Scan Before and After Radiation Therapy for the Detection of Intracranial Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1008; NCI-2021-03217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1008 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-09

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (advanced MRI) (Experimental): Patients undergo conventional and advanced MRI over 60 minutes within 14 days before the start of scheduled brain radiation treatment. Patients then undergo 7 additional MRI over 60 minutes each between 4-16 weeks apart. Patients may receive gadolinium and/or iopamidol during MRI scans.
  Interventions: Procedure: Advanced Magnetic Resonance Imaging; Procedure: Conventional Magnetic Resonance Imaging; Drug: Gadolinium-Chelate; Drug: Iopamidol

INTERVENTIONS:
Procedure: Advanced Magnetic Resonance Imaging — Undergo advanced MRI
  Other Names: AMRI
Procedure: Conventional Magnetic Resonance Imaging — Undergo conventional MRI
  Other Names: Conventional MRI
Drug: Gadolinium-Chelate — Contrast agent
  Other Names: Gadolinium Coordination Complex; Gadolinium-based Contrast Agent; Gadolinium-Chelant Complex
Drug: Iopamidol — Contrast agent
  Other Names: Isovue; Niopam; Solutrast

SUMMARY:
This clinical trial studies the different types of investigational imaging techniques called sequences during magnetic resonance imaging (MRI) of the head before and after radiation therapy in patients with cancer that has spread to the brain (intracranial metastases). This clinical trial also compares these new techniques with standard MRI imaging to see if sequences provide better images. Diagnostic procedures, such as MRI, may help find and diagnose solid organ cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conspicuity:

Ia. To assess the conspicuity of idealized T1 and T2 imaging at detecting brain metastases at baseline. (Quantitative MRI) Ib. To assess the conspicuity (CNR) of chemical exchange saturation transfer (CEST) imaging at detecting brain metastases at baseline. (CEST MRI) Ic. To assess the conspicuity (CNR) of advances in difference equations (Adv Diff) at detecting brain metastases at baseline. (Multiple B Value Diffusion Imaging [Adv Diff]) Id. To assess the conspicuity of gradient- and spin-echo (GESE) dynamic susceptibility contrast (DSC) and standard Gradient Echo (GE) DSC at detecting brain metastases at baseline. (GESE DSC perfusion imaging)

SECONDARY OBJECTIVES:

I. Conspicuity:

Ia. To assess the conspicuity of T2 imaging at detecting brain metastases on a per-patient basis at follow-up scans and on a per-lesion basis at baseline and at follow-up time points. (Quantitative MRI) Ib. To assess the conspicuity (CNR) of CEST imaging at detecting brain metastases on a per-patient basis at follow-up scans and on a per-lesion basis at baseline and at follow-up time points. (CEST MRI) Ic. To assess the conspicuity (CNR) of Adv Diff at detecting brain metastases on a per-patient basis at follow-up scans and on a per-lesion basis at baseline and at follow-up time points. (Multiple B Value Diffusion Imaging [Adv Diff]) Id. To assess the conspicuity of GESE DSC and standard Gradient Echo (GE) DSC at detecting brain metastases on a per-patient basis at follow-up scans and on a per-lesion basis at baseline and at follow-up time points. (GESE DSC perfusion imaging) II. Treatment response. IIa. To assess the trend of idealized quantitative T1 and T2 values of brain metastases compared to normal brain parenchyma following treatment with stereotactic radiosurgery. (Quantitative MRI) IIb. To assess the ability of CEST imaging to differentiate radiation necrosis from progressive disease in brain metastases following stereotactic radiosurgery. (CEST MRI) IIc. To assess whether Adv Diff can differentiate radiation necrosis from progressive disease in brain metastases following stereotactic radiosurgery. (Multiple B Value Diffusion Imaging [Adv Diff]) IId. To assess whether GESE DSC improves differentiation of radiation necrosis from progressive disease in brain metastases following stereotactic radiosurgery compared to standard GE DSC. (GESE DSC perfusion imaging) IIe. To assess the ability of Adv arterial spin labeling (ASL) to differentiate radiation necrosis from progressive disease in brain metastases following stereotactic radiosurgery. (Multiple inversion time [TI] ASL "Adv ASL" perfusion)

OUTLINE:

Patients undergo conventional and advanced MRI scans over 60 minutes within 14 days before the start of scheduled brain radiation treatment. Patients then undergo 7 additional MRI scans over 60 minutes each between 4-16 weeks apart. Patients may receive gadolinium and/or iopamidol during MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* An adult patient with pathology-proven solid organ cancer
* MRI of the brain with contrast, positive for at least one intra-axial metastatic lesion greater than 5 mm
* Planned treatment with stereotactic radiation

Exclusion Criteria:

* Contraindication to MR imaging
* Known allergy to gadolinium-based contrast agents
* Renal failure as defined by a glomerular filtration rate (GFR) less than 30 or the use of hemodialysis
* Pregnant
* Patients less than 18 years of age will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with brain metastases were scanned on a dual-energy CT scanner following iohexol injection at four different time points
Groups:
- Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery: Single Arm
Period: Overall Study
Arm/Group | Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Contrast to Noise Ratio
Description: Contrast enhancement compared to baseline and normalized to background noise
Time Frame: Participants enrolled in the study were followed for variable amounts of times (up to 2 years and 4 months) from the date of their enrollment and baseline imaging
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery
Number analyzed (Participants) | 15
Ratio | 3.2 (1.1)
Statistical Analysis 1: Comparison: Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery; Test type: Other; p < 0.05, Statistical Significance

ADVERSE EVENTS:
Time Frame: Participants enrolled in the study were followed for variable amounts of times (up to 2 years and 4 months) from the date of their enrollment and baseline imaging.
Arm/Group | Advanced MRI for Intracranial Metastasis Treated With Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT04870645/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT04870645/ICF_001.pdf